CLINICAL TRIAL: NCT02994199
Title: Use of Adapted Controllers for Active Video Gaming (Interactive Exercise and Recreation Technologies and Exercise Physiology Benefiting People With Disabilities)
Brief Title: Use of Adapted Controllers for Active Video Gaming in People With Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laurie A Malone, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: F150909002
Record Dates: First submitted 2016-12-06; First posted 2016-12-15 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Physical Disability
Keywords: Active video gaming; Energy expenditure
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active video gaming (Experimental): Participants will engage in active video game play.
  Interventions: Other: Active video gaming

INTERVENTIONS:
Other: Active video gaming — Participants will engage in active video game play using two off-the-shelf (OTS) and two adapted controllers using the Wii gaming console. Controllers are: OTS balance board, OTS gaming mat, Adapted balance board, Adapted gaming mat.

SUMMARY:
The purpose of this study is to compare the effectiveness of off-the-shelf (OTS) and adapted game controllers on quality of game play, enjoyment, and energy expenditure during active video gaming in persons with mobility impairments. The controllers to be evaluated include off-the-shelf and adapted gaming mats and off-the-shelf and adapted Wii Fit balance boards.

DETAILED DESCRIPTION:
Previous studies have shown that individuals with disabilities have lower levels of physical activity and fitness and higher levels of obesity compared to their non-disabled peers. Research has also shown that engaging this population in physical activity can be extremely challenging due to physical impairments associated with their disability, as well as fewer opportunities to participate.

Active video games (AVG), also known as exergames, are a category of video games that require much more body motion for successful play than the traditional pushbutton or joystick actions. The recent introduction of motion controlled AVGs allow a much greater variety of physical activity to be part of play. These games hold promise for promoting higher levels of energy expenditure, weight management and fitness. However, many current AVGs are inaccessible or offer limited play options for individuals who are unable to stand, have balance issues, poor motor control, or cannot use their lower body to perform game activities. Making AVGs accessible to people with disabilities offers an innovative approach to overcoming various barriers to participation in beneficial physical activity.

A recent publication by Dr. Rimmer in the Physical Medicine and Rehabilitation journal examining the use of AVGs as a means to increase energy expenditure in non-ambulatory young adults with disabilities suggested that clinically significant increases in energy expenditure could be achieved with AVGs.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants must have a confirmed diagnosis of lower extremity mobility disability (e.g., spina bifida, cerebral palsy, muscular dystrophy,1 year post spinal cord injury, multiple sclerosis, stroke, or limb loss) with partial or full use of upper extremities and use of an assistive device (manual wheelchair, walker, crutches, or canes) for balance and/or mobility or should have gait deviation.
* Participants must be between the ages of 10 and 60 yrs, and not weigh more than 350 pounds.

Exclusion Criteria:

* Unstable cardiovascular conditions as identified by their physician.
* Weight over 350 pounds
* Visual impairment that interferes with playing video games

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Energy expenditure (ml/kg/min) | Visit 1: baseline measurement at rest
  Measured using a portable metabolic system
Energy expenditure (ml/kg/min) | Visit 2: during game play
  Measured using a portable metabolic system
Energy expenditure (ml/kg/min) | Visit 3: during game play
  Measured using a portable metabolic system

SECONDARY OUTCOMES:
Enjoyment | Visit 2: following first game set
  Participants will complete the Physical Activity Enjoyment Scale (PACES)
Enjoyment | Visit 2: following second game set
  Participants will complete the Physical Activity Enjoyment Scale (PACES)
Enjoyment | Visit 3: following first game set
  Participants will complete the Physical Activity Enjoyment Scale (PACES)
Enjoyment | Visit 3: following second game set
  Participants will complete the Physical Activity Enjoyment Scale (PACES)
Quality of game play | Visit 2: following first game set
  Subjective evaluation by the tester: degree of general game manipulation in comparison to able-bodied gamer; Likert scale 0 (unable) to 5 (excellent)
Quality of game play | Visit 2: following second game set
  Subjective evaluation by the tester: degree of general game manipulation in comparison to able-bodied gamer; Likert scale 0 (unable) to 5 (excellent)
Quality of game play | Visit 3: following first game set
  Subjective evaluation by the tester: degree of general game manipulation in comparison to able-bodied gamer; Likert scale 0 (unable) to 5 (excellent)
Quality of game play | Visit 3: following second game set
  Subjective evaluation by the tester: degree of general game manipulation in comparison to able-bodied gamer; Likert scale 0 (unable) to 5 (excellent)
Controller usability | At the completion of Visit 2
  Participants will complete the System Usability Scale
Controller usability | At the completion of Visit 3
  Participants will complete the System Usability Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Padalabalanarayanan, MS, Study Director — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malone LA, Padalabalanarayanan S, McCroskey J, Thirumalai M. Assessment of Active Video Gaming Using Adapted Controllers by Individuals With Physical Disabilities: A Protocol. JMIR Res Protoc. 2017 Jun 16;6(6):e116. doi: 10.2196/resprot.7621. PMID 28623186
- [Result] Malone LA, Thirumalai M, Padalabalanarayanan S, Neal WN, Bowman S, Mehta T. Energy Expenditure and Enjoyment During Active Video Gaming Using an Adapted Wii Fit Balance Board in Adults with Physical Disabilities: Observational Study. JMIR Serious Games. 2019 Feb 1;7(1):e11326. doi: 10.2196/11326. PMID 30707098
- [Result] Thirumalai M, Kirkland WB, Misko SR, Padalabalanarayanan S, Malone LA. Adapting the Wii Fit Balance Board to Enable Active Video Game Play by Wheelchair Users: User-Centered Design and Usability Evaluation. JMIR Rehabil Assist Technol. 2018 Mar 6;5(1):e2. doi: 10.2196/rehab.8003. PMID 29510972
- [Result] Malone LA, Davlyatov GK, Padalabalanarayanan S, Thirumalai M. Active Video Gaming Using an Adapted Gaming Mat in Youth and Adults With Physical Disabilities: Observational Study. JMIR Serious Games. 2021 Aug 26;9(3):e30672. doi: 10.2196/30672. PMID 34435962